CLINICAL TRIAL: NCT06779396
Title: Pre-emptive Scalp Infiltration with Triamcinolone Acetonide Plus Ropivacaine for Post-Craniotomy Pain in Children
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY 2018-066-02-4
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Pain; Postoperative Children
Keywords: Postoperative Pain; Pre-emptive Scalp Infiltration; Triamcinolone Acetonide
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: The triamcinolone acetonide plus ropivacaine group (Experimental): Patients in the triamcinolone acetonide plus ropivacaine group will receive a peri-incisional scalp infiltration with 0.2% ropivacaine(40mg) and 4 mg of triamcinolone acetonide and normal saline miscible liquids.
  Interventions: Drug: The triamcinolone acetonide plus ropivacaine group
- Active Comparator: The ropivacaine group (Active Comparator): Patients in the ropivacaine group will receive a peri-incisional scalp infiltration 0.2% ropivacaine(40mg)
  Interventions: Drug: The ropivacaine group

INTERVENTIONS:
Drug: The triamcinolone acetonide plus ropivacaine group — The solution prepared comprised a mixture of 20mL of 0.2% ropivacaine(40mg) with 4 mg of triamcinolone acetonide. The assigned solution will be injected subcutaneously by surgeons along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigators.
  Arms: Experimental: The triamcinolone acetonide plus ropivacaine group
Drug: The ropivacaine group — The local infiltration solution containing 20mg of 1% ropivacaine. The total volume is 20 ml. The assigned solution will be injected subcutaneously by surgeons along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigators.
  Arms: Active Comparator: The ropivacaine group

SUMMARY:
At present, pediatric postoperative analgesia has not been fully understood and controlled, particularly craniotomy surgery. On the one hand, professional evaluation of postoperative pain for young children is difficult; on the other hand, the particularity of craniotomy adds (such as consciousness obstacle, sleepiness, et al) disturbance to the pain assessment in children. Although opioids administration is regarded as the first-line analgesic for post-craniotomy pain management, it may be associated with delayed awakening, respiratory depression, hypercarbia and it may interfere with the neurologic examination. For the avoidance of side-effects of systemic opioids, local anesthetics administered around the incision have been performed clinically. However, some studies revealed that the analgesic effect of local anesthetics was unsatisfactory due to its short pain relief duration, steroid as adjuvant can enhance postoperative analgesia and prolong postoperative analgesia time. As is reported that postoperative pain of craniotomy is mainly caused by skin incision and reflection of muscles, preventing the liberation of inflammatory mediators around the incision seems to be more effective than simply blocking nerve conduction.However, there has not been reported about local application of triamcinolone acetonide on scalp infiltration. Thus, the investigators suppose that pre-emptive scalp infiltration with steroid (triamcinolone acetonide) plus local anesthetic (ropivacaine) could relieve postoperative pain after craniotomy in children.

ELIGIBILITY:
Inclusion Criteria:

-(1) Age 2 to 12 years. (2) American Society of Anesthesiologists (ASA) physical status I or II. (3)Participates with an anticipated fully recovery within 2 hours postoperatively.

(4)Informed consent by parent(s) and/or legal guardian.

Exclusion Criteria:

- (1) Allergy to local anesthetics. (2) Pediatric patients aged>12 or <2 years. (3) Under medication with analgesic drugs. (4) Psychiatric disorders. (5) Uncontrolled epilepsy. (6) Chronic headache. (7) Peri-incisional infection. (8) Coagulopathy or bleeding disorder. (9) Patients who are expected to remain intubated and mechanical ventilation after surgery.

(10) Emergency craniotomies. (11) Patients with cardiac insufficiency or severe kidney or liver diseases. (12) Patients whose authorized surrogates are unwilling to participate in the study

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
the Faces, Legs, Activity, Cry, Consolability (FLACC) scale | At 24 hours after the operation
  Postoperative pain will be estimated by usingthe Faces, Legs, Activity, Cry, Consolability (FLACC) scale score at 24 hours postoperatively.

SECONDARY OUTCOMES:
the Faces, Legs, Activity, Cry, Consolability (FLACC) scale | At 2 hours, 4 hours, 8 hours, 48 hours, 72 hours, 1 week after surgery
  Postoperative pain will be estimated by using the Faces, Legs, Activity, Cry, Consolability (FLACC) scale
Duration of analgesia | Within 48 hours after the operation
  the time to the first postoperative analgesic request
The occurrence of postoperative nausea and vomiting (PONV) | At 2 hours, 4 hours, 8 hours, 24 hours after surgery
  PONV will be rated by participants as: 0, absent; 1, nausea not requiring treatment; 2, nausea requiring treatment; and 3, vomiting.
Incisional related adverse events | Approximately 1 weeks after the operation
  Incisional related adverse events Including delayed incisional healing, incisional infection, intracranial infection, scar healing.
The occurrence of the Adverse events (AEs) and serious adverse events (SAEs) | Within 1 weeks after the operation
  An AE was defined as any untoward medical occurrence. An SAE included death, immediately life-threatening conditions, coma, in-patient hospitalisation or prolongation of existing hospitalisation.
Patient satisfactory scale (PSS) | At 2 hours, 4 hours, 8 hours, 48 hours, 72 hours, 1 week after surgery
  0 for unsatisfactory, and 10 for very satisfied
The total consumption of opioids during the operation | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.